CLINICAL TRIAL: NCT00310908
Title: Efficacy of Tramadol Hcl in the Treatment of Renal Colic
Brief Title: Comparison Between Tramadol Hcl and Other Analgesics in the Treatment of Renal Colic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Grumental (Unknown)
Responsible Party: Ruth Stalnikowicz, Hadassah Medical Organization
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1234567-HMO-CTIL
Record Dates: First submitted 2006-04-04; First posted 2006-04-05 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2006-09

CONDITIONS: Renal Calculus
Keywords: Renal; Colic; Calculi; Treatment
MeSH Terms: conditions — Kidney Calculi; Colic; Calculi | interventions — Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tramadol Hcl — Active Comparator

SUMMARY:
The purpose of this study is to determine whether Tramadol Hcl is as effective as Voltaren a non-steroidal antiinflammatory drug, and Dipyrone in amelioration of the pain caused by acute renal colic.

DETAILED DESCRIPTION:
Renal stones is a common condition affecting up to 1% of the american population. The main symptom is renal colic. Acute treatment is based on the administration of analgesics mainly those belonging to non-steroidal antiinflammatory drugs (NSAIDs). Tramadol is an analgesic of the opioid class of analgesics (i.e morphine) and it is considered to cause less side effects with more or less the same analgesic potency. In the present study the analgesic effect of intramuscular Tramadol will be compared with Voltaren (NSAID)in patients attending the Emergency Department (ED) for acute renal colic (Stage I). Most of these patients will not pass their stone during their visit to the ED and they are prone to develop another attack of renal colic.In the second phase of the study (Stage II)patients who improved, and are ready to go home, will be enrolled to get Dipyrone or Tramadol orally for the prevention of further pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of acute renal colic (Stage I)
* Patients with diagnosed renal colic who might need prevention of pain and are able to swallow medicines (Stage II)

Exclusion Criteria:

* Patients with known hypersensitivity to the study drugs
* Pregnancy or lactation
* Known renal failure or hepatic disease
* Concommitant drug use which could adversely affect patient's outcome (oral anticoagulant, MAO inhibitors)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pain improvement according to VAS score at 30, 60 and 120 minutes(Stage I) | 30, 60, 120 minutes
Need for rescue medication at 30 minutes (Stage I) | 30 minutes
Pain improvement according to VAS score at 24 and 48 hrs (Stage II) | 24 and 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Stalnikowicz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Ukhal' MI, Melenevskii DA. [Using prostaglandin inhibitor dicloberl in patients with ureteral calculi]. Lik Sprava. 2004 Mar;(2):76-8. Russian. PMID 15208882